CLINICAL TRIAL: NCT01530243
Title: Phase One of Study on Urinary Stent Complications and Treatment
Brief Title: The Effect of Terazosin and Tolterodine on Ureteral Stent Related Symptoms
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Urmia University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UUNRC 01
Record Dates: First submitted 2012-01-18; First posted 2012-02-09 (Estimated); Results first posted 2015-03-02 (Estimated); Last update posted 2015-03-02 (Estimated); Status verified 2015-02

CONDITIONS: Disorder of Urinary Stent
MeSH Terms: interventions — Terazosin; Tolterodine Tartrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Terazosin (Active Comparator)
  Interventions: Drug: Terazosine
- Tolterodine (Active Comparator)
  Interventions: Drug: Tolterodine
- Tolterodine + Terazosin (Active Comparator)
  Interventions: Drug: Tolterodine + Terazosin

INTERVENTIONS:
Drug: Placebo — same as tolterodine and terazosin dose
  Other Names: Group 1
  Arms: Placebo
Drug: Terazosine — 2 mg BID
  Other Names: Group 2
  Arms: Terazosin
Drug: Tolterodine — 2 mg daily
  Other Names: Group 3
  Arms: Tolterodine
Drug: Tolterodine + Terazosin — 2mg daily and 2mg BID
  Other Names: Group 4
  Arms: Tolterodine + Terazosin

SUMMARY:
The aim of the investigators study is to evaluate whether alpha-blockers such as terazosin and anti-cholinergics such as tolterodine can be relieve the DJ-stent related symptoms.

DETAILED DESCRIPTION:
Ureteral stent (US) has been as essential tool in the urologist's surgeries and is useful instruments that its indications increase due to new stent technologies and improvement of patient's comfort.

US associated with discomfort complications that include lower urinary tract symptoms (LUTS) as frequency, urgency, dysuria, incomplete emptying, flanks and suprapubic's pain, incontinence, hematuria, movement of stent, infection and encrustation of stent. US related symptoms are as same as LUTS due to benign prostate hyperplasia and overactive bladder which relieve with alpha-blockers and anticholinergic. The purpose of our study is to investigate the effect of terazosin and tolterodine lonely and together in comparison of placebo on US related symptoms.

The investigators study will be done prospectively. The patients who underwent indwelling Double-j stent distributed into four groups: 1)receive placebo 2)receive terazosin 2mg twice 3)receive tolterodine 2mg daily 4) receive terazosin 2mg twice and tolterodine 2mg daily. All of the patients receive prophylactic antibiotic and on demand analgesic. After entrance to study, they fulfill the International Prostatic Symptoms Score (IPSS) and Visual Analog Scale (VAS) on the before indwelling US, two weeks after indwelling US and US removal time, then the investigators will evaluate the drug's effect on US related symptoms.

ELIGIBILITY:
Inclusion Criteria:

If a patient does not meet any exclusion criteria and to be undergone double-J stent indwelling.

Exclusion Criteria:

1. Prior history of pelvic surgery
2. Prior history of Transurethral Resection of the either Prostate or Bladder Tumor
3. Benign prostate hyperplasia
4. Recent or recurrent urinary tract infection
5. Chronic medication with beta-blockers or Anti-cholinergic
6. Pregnancy
7. Prostatitis
8. Prostate cancer
9. Bilateral ureteroscopy or ureteral stenting
10. Age < 18 and > 55
11. Stone size > 20 mm
12. Diabetes
13. Bladder Outlet Obstruction

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2012-01; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ali Tehranchi, Urologist, Study Chair — Urology department; Yousef Rezaei, M.D, Principal Investigator — Urmia University of Medical Sciences
Locations (1):
- Imam Khomeini Hospital, Urmia, Azerbaijan-gharbi, Iran

REFERENCES:
- [Background] Tehranchi A, Rezaei Y, Khalkhali H, Rezaei M. Effects of terazosin and tolterodine on ureteral stent related symptoms: a double-blind placebo-controlled randomized clinical trial. Int Braz J Urol. 2013 Nov-Dec;39(6):832-40. doi: 10.1590/S1677-5538.IBJU.2013.06.09. PMID 24456787

RESULTS

PARTICIPANT FLOW:
Groups:
- Terazosin: Terazosin: 2 mg BID
Period: Overall Study
Arm/Group | Placebo | Terazosin | Tolterodine | Tolterodine + Terazosin
Started | 26 | 26 | 26 | 26
Completed | 24 | 23 | 23 | 24
Not Completed | 2 | 3 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Terazosin | Tolterodine | Tolterodine + Terazosin | Total
Number analyzed (Participants) | 24 | 23 | 23 | 24 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.37 (9.58) | 38.35 (9.23) | 37.04 (9.04) | 35.75 (9.38) | 36.53 (9.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 4 | 5 | 19
  Male | 21 | 16 | 19 | 19 | 75
Region of Enrollment [Number; unit: participants]
  Iran, Islamic Republic of | 24 | 23 | 23 | 24 | 94

OUTCOME MEASURES:

1. Primary Outcome: Lower Urinary Tract Symptoms (LUTS)
Description: LUTS was evaluated using the International Prostate Symptom Score (IPSS) questionnaire perioperatively. The IPSS constitutes of seven questions assigned score from 0 to 5 to evaluate the severity of LUTS in patients. Total scoring of IPSS ranges from 0 to 35, asymptomatic to very symptomatic. The more the score on scale is, the worse the outcome is.Therefore, the higher values represent worse outcomes.
Time Frame: Expected average of 2 weeks
Population: The more the score on scale is, the worse the outcome is.Therefore, the higher values represent worse outcomes.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Terazosin | Tolterodine | Tolterodine + Terazosin
Number analyzed (Participants) | 24 | 23 | 23 | 24
units on a scale | 11.12 (7.84) | 4.39 (6.03) | 7.21 (6.57) | 5.58 (4.82)

2. Secondary Outcome: Quality of Life
Description: The Quality of life of patients was evaluated using single question in IPSS questionnaire in which each of patients received scoring from 0 to 6. The higher values represent the worse quality of life.
Time Frame: Expected 2 weeks later
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Terazosin | Tolterodine | Tolterodine + Terazosin
Number analyzed (Participants) | 24 | 23 | 23 | 24
units on a scale | 3.37 (2.16) | 2 (2.25) | 2.30 (1.89) | 0.95 (1.12)

3. Other Pre Specified Outcome: Pain
Description: The visual analogue scale (VAS) was used to evaluate the pain at the time of voiding. This VAS scoring ranges from 0 to 10. The higher values represent worse outcomes, having more pain.
Time Frame: Expected 2 weeks later
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Terazosin | Tolterodine | Tolterodine + Terazosin
Number analyzed (Participants) | 24 | 23 | 23 | 24
units on a scale | 4.16 (3.59) | 3.21 (4.14) | 1.34 (2.60) | 1.37 (2.56)

ADVERSE EVENTS:
Arm/Group | Placebo | Terazosin | Tolterodine | Tolterodine + Terazosin
Serious Adverse Events (participants affected / at risk) | 2/24 | 4/23 | 1/23 | 6/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/23 | 0/23 | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=24) | Terazosin (N=23) | Tolterodine (N=23) | Tolterodine + Terazosin (N=24)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 4 (4) | 1 (1) | 6 (6)

LIMITATIONS AND CAVEATS:
Applying stents with the same size and length

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No